CLINICAL TRIAL: NCT00001975
Title: Cutaneous Tumorigenesis in Patients With Tuberous Sclerosis
Brief Title: Study of Skin Tumors in Tuberous Sclerosis
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000051; 00-H-0051
Record Dates: First submitted 2000-01-20; First posted 2000-01-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-16

CONDITIONS: Tuberous Sclerosis
Keywords: Skin Biopsy; Familial Tumor Syndrome; Cell Growth; Loss of Heterozygosity; Cytokines; Natural History; Tuberous Sclerosis
MeSH Terms: conditions — Tuberous Sclerosis; Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients will be those already diagnosed with TSC (definite or possible)

SUMMARY:
Tuberous sclerosis is a rare, hereditary disease in which patients develop multiple tumors. Although not cancerous, the tumors can affect various organs, including the heart, lungs, kidneys, skin, and central nervous system, with serious medical consequences. The severity of disease varies greatly among patients, from barely detectable to fatal. This study will investigate what causes skin tumors to develop in patients with this disease.

Patients with tuberous sclerosis 18 years and older may enroll in this study. Participants will undergo a medical history and thorough skin examination by a dermatologist. Those with skin tumors will be asked to undergo biopsy (tissue removal) of up to eight lesions, under a local anesthetic, for research purposes. The biopsies will all be done the same day. The tissue samples will be used for: examination of genetic changes, measurement of certain proteins and other substances, and growing in culture to study the genetics of tuberous sclerosis.

DETAILED DESCRIPTION:
Patients with tuberous sclerosis develop benign cutaneous tumors that are typically multiple in number and location. These tumors include facial angiofibromas, forehead plaques, shagreen patches, periungual fibromas, and gingival fibromas. The tumors are permanent, slow growing, and often disfiguring. The purpose of this study is to elucidate the molecular basis for these tumors. Specifically, we plan to identify the genetically altered cells in these hamartomatous lesions, and to quantify factors (e.g. cytokines) produced by these cells which induce the growth of these tumors. To accomplish this, we plan to obtain samples of these cutaneous tumors, to test tumor DNA for loss of heterozygosity, and to measure RNA and protein expression levels.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be those already diagnosed with TSC (definite, probable, or possible) based on clinical criteria and/or genetic testing, and ranging in age from 18 to 90 years old.

The clinical features of TSC considered of major significance are: facial angiofibromas or forehead plaque, nontraumatic periungual fibromas, three or more hypomelanotic macules, shagreen patch, multiple retinal nodular hamartomas, cortical tuber, subependymal nodule, subependymal giant cell astrocytoma, cardiac rhabdomyoma, lymphangioleiomyomatosis, and renal angiomyolipoma.

The minor features of TSC are: multiple randomly distributed pits in dental enamel, hamartomatous rectal polyps, bone cysts, cerebral white matter radial migration lines, gingival fibromas, nonrenal hamartoma, retinal achromic patch, confetti skin lesions, and multiple renal cysts (5). Definite TSC is diagnosed by the presence of two major features or one major feature plus two minor features. Probable TSC is diagnosed by the presence of one major feature and one minor feature. Possible TSC is diagnosed by the presence of either one major feature or two or more minor features. Patients will not be preselected for skin lesions, but about 80% of patients with TSC are expected to have skin lesions.

EXCLUSION CRITERIA:

Inability to give informed consent.

Tendency to keloid formation.

Allergy to anesthetics.

Bleeding abnormality.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be those already diagnosed with TSC (definite or possible) based on clinical criteria and/or genetic testing, and ranging in age from 18 to 90 years old.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2000-01-26 (Actual)

PRIMARY OUTCOMES:
1.Identify the tumor cells in cutaneous and mucosal tumors in patients with TSC through LOH studies on microdissected cell populations | ongoing
  natural history

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a new requirement and the sharing of IPD is not discussed in the protocol.

REFERENCES:
- [Background] Kwiatkowski DJ, Short MP. Tuberous sclerosis. Arch Dermatol. 1994 Mar;130(3):348-54. PMID 8129414
- [Background] Weiner DM, Ewalt DH, Roach ES, Hensle TW. The tuberous sclerosis complex: a comprehensive review. J Am Coll Surg. 1998 Nov;187(5):548-61. doi: 10.1016/s1072-7515(98)00239-7. No abstract available. PMID 9809574
- [Background] Webb DW, Clarke A, Fryer A, Osborne JP. The cutaneous features of tuberous sclerosis: a population study. Br J Dermatol. 1996 Jul;135(1):1-5. PMID 8776349
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-H-0051.html